CLINICAL TRIAL: NCT04481529
Title: Study of the COVID-19 Serological Status of Hospital Staff Working or Not in the COVID-19 Sector in 3 French Regions Facing the COVID-19 Epidemic With Varying Degrees of Intensity
Brief Title: COVID-19 Serological Status of Hospital Staff Working or Not in the COVID-19 Sector
Acronym: SEROCO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI20_0049/SEROCO
Record Dates: First submitted 2020-07-20; First posted 2020-07-22 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-11

CONDITIONS: Infection Viral
MeSH Terms: conditions — Virus Diseases | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Health Questionnaire — Completion of a short questionnaire noting the result of the serology and looking for elements in favor of exposure to the virus, whether professional or extra-professional.

SUMMARY:
Hospital staff, on the front line in the COVID-19 crisis, have many questions about the risk that they have been infected with this potentially fatal virus. These questions of course primarily concern caregivers working in sectors dedicated to COVID-19 patients, whether they are resuscitating or not, but also those in non-COVID-19 sectors, or even staff without direct contact with patients. In addition, depending on the suddenness and intensity of this "COVID-19 wave", these personnel have been more or less trained and sometimes exposed due to the dire lack of protective equipment. In some countries such as Great Britain, this has resulted in significant absenteeism, a source of deepening the shortage of caregivers.

This proportion of contaminated caregivers has not been evaluated on the whole of French territory. Studies from other countries suggest figures ranging from 1.5% in China to 20% in Italy. It is therefore impossible to rely on such variable data to have a reliable estimate.

Since june 2020, all staff in French health establishments could benefit a serological test.

Thus, in this epidemiological study, we propose to rely on this institutional serological screening to describe the link between seroconversion of hospital staff, regional intensity of the epidemic, and sectors of activity (COVID-19 sectors, non-COVID-19 caregivers , non-COVID-19 non-caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Hospital staff from Argenteuil, Belfort, Dijon and Limoges hospitals.
* Age ≥ 18 years old
* Participation agreement

Exclusion Criteria:

* Protected persons
* Refusal of participation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hospital staff
Sampling Method: Non-Probability Sample
Enrollment: 1576 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with a COVID-19 seroconversion | through study completion, an average of 5 month
  Number of subjects with a COVID-19 seroconversion fixed by the presence of IgG + in serology according to the service (COVID19 +, COVID19- caregiver, COVID- non-caregiver).

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CH Argenteuil - Service de Réanimation, Argenteuil
  - Ch Belfort, Belfort
  - CHU Dijon - Serve de Réanimation, Dijon
  - CHU de Limoges, Limoges